CLINICAL TRIAL: NCT06183593
Title: Accuracy in the Evaluation of Brain Response to Mechanical and Radiofrequency Stimuli in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Collaborators: Medical School Hamburg (Other)
Responsible Party: Principal Investigator, Christian Mista, Principal Investigator, National Council of Scientific and Technical Research, Argentina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IS004486
Record Dates: First submitted 2023-12-14; First posted 2023-12-27 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Brain Response Evoked by Radiofrequency Stimuli in Humans; Brain Response Evoked by Pinprick Stimuli in Humans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency-evoked potentials (RFEPs) (Experimental): The application of RF stimuli will be carried out using an adapted electrocoagulation device (ECD). These devices have several types of applicators, depending on the type of stimulation to be performed. In the bipolar mode, the applicator consists of a small clamp whose tips constitute the active and return electrodes, and the electric current flows only through the tissue captured between the two tips of the clamp. In the unipolar mode, the active electrode is an interchangeable tip with a variable surface (resembling for example a blade or a needle), and the return electrode is a metal plate in contact with another part of the volunteer's body. In this case, the current also flows from the active electrode to the return electrode, but over a considerably longer path. In both cases the physiological effect is similar: the stimulation elicits superficial, localized and limited heating of the tissue in the vicinity of the active electrode.
  Interventions: Other: Radiofrequency application
- Pinprick evoked potentials (Experimental): An automatic stimulator with a section of approximately 0.35 mm in diameter and with a blunt tip was developed to apply this type of stimulus. This stimulator has a calibrated spring, which allows force to be gradually applied, while providing a safety margin to avoid accidents during tests. This allows two types of measurements to be made depending on the speed with which the stimulus is applied.
  Interventions: Other: Pinprick stimuli

INTERVENTIONS:
Other: Radiofrequency application — Radiofrequency stimuli will be applied at pain threshold intensity. Arm and leg will be stimulated.
  Arms: Radiofrequency-evoked potentials (RFEPs)
Other: Pinprick stimuli — Pinprick stimuli will be administered at varying speeds and forces using an automated device
  Arms: Pinprick evoked potentials

SUMMARY:
Under normal conditions, pain arises as a consequence of the activation of nociceptive afferents (small fibers) by an external stimulus with sufficient intensity to potentially cause tissue damage. This peripheral activation is processed as perception of pain by the central nervous system. In order to reliably evaluate the state of the nociceptive system in both clinical and experimental settings, standardized tests are essential. Quantitative sensory testing (QST) is a set of tests used to measure the intensity of a stimulus that produces a specific sensory perception in a subject. For example, if we gradually apply pressure, the point where the sensation changes from pressure to pain is called the pressure pain threshold. This type of test can be performed with different types of stimuli, including hot and cold stimuli or mechanical stimuli. Although these tests have been shown as reliable in healthy volunteers and pain patients, they are subjective in their nature, since they are based on a conscious evaluation of tested subjects. Likewise, these measures show substantial variability due to differences in the application of the tests by individual examinators. In short, even though the method is quantitative, its methodological characteristics make it subjective and dependent on both the operator and the subject under study. Moreover, contrasting results have been recently found regarding the measurement variability when repeating the QST at intervals of days. Thus, it is essential to investigate and develop new QST alternatives to obtain objective markers that may potentially contribute to the understanding of the mechanisms behind chronic pain conditions.

DETAILED DESCRIPTION:
Under normal conditions, pain arises as a consequence of the activation of nociceptive afferents (small fibers) by an external stimulus with sufficient intensity to potentially cause tissue damage. This peripheral activation is processed as perception of pain by the central nervous system. In order to reliably evaluate the state of the nociceptive system in both clinical and experimental settings, standardized tests are essential. Quantitative sensory testing (QST) is a set of tests used to measure the intensity of a stimulus that produces a specific sensory perception in a subject. For example, if we gradually apply pressure, the point where the sensation changes from pressure to pain is called the pressure pain threshold. This type of test can be performed with different types of stimuli, including hot and cold stimuli or mechanical stimuli. Although these tests have been shown as reliable in healthy volunteers and pain patients, they are subjective in their nature, since they are based on a conscious evaluation of tested subjects. Likewise, these measures show substantial variability due to differences in the application of the tests by individual examinators. In short, even though the method is quantitative, its methodological characteristics make it subjective and dependent on both the operator and the subject under study. Moreover, contrasting results have been recently found regarding the measurement variability when repeating the QST at intervals of days. Thus, it is essential to investigate and develop new QST alternatives to obtain objective markers that may potentially contribute to the understanding of the mechanisms behind chronic pain conditions.

In this regard, evoked potentials (EP) measured by electroencephalography (EEG) are the most commonly used objective alternative for the functional evaluation of small fibers and the spinothalamic tract. Nociceptive EPs can be induced with various stimulation modalities, including lasers (LEP), contact heat (CHEP) and cold (CCEP), intradermal electrical stimulation (IEEP), and mechanical needling (PEP), and each modality has its own advantages and disadvantages. Recently, a novel type of EP has been proposed that is evoked by electrical stimulation in the range of 200 kHz to 3.3 MHz, that is, in the radio frequency (RF) spectrum. At such high frequencies, the nerves and muscles can no longer be electrically excited, and the physiological effects are generated exclusively due to the heating of the tissue. In strictly physiological terms, RF electrical stimuli are similar to those generated by contact heat. Importantly, non-ablative RF technology is safe, relatively inexpensive, and in widespread use in clinics (Beasley & Weiss, 2014; Lolis & Goldberg, 2012)- Therefore, the use of RF stimulation could significantly increase the accessibility of EPs as a reference electrophysiological tool for the evaluation of the state of the nociceptive system.

Another attractive alternative to subjective evaluation is the EP elicited by sharp mechanical stimuli (pinprick). A device that applies this type of stimulus has recently been developed. It uses a stimulator with a tip similar to that of a blunt needle, which allows obtaining brain responses synchronized with the stimulus and evaluating the state of the spino-thalamic-cortical mechanical sensory conduction pathways. At the Faculty of Engineering of the National University of Entre Ríos (FI-UNER), a prototype was developed that allows it to be carried out in an automated manner, which allows to reduce the uncertainty derived from human subjectivity.

In the proposed protocol, the precision of the brain response to RF and mechanical sharp stimuli will be evaluated in two experimental settings. We plan to assess the effect of stimulation intensity on signal parameters, such as EP latency and amplitude. Furthermore, the relationship of these parameters with psychophysical results (questionnaires) and heat thresholds will be explored to investigate the relationship between these variables.

ELIGIBILITY:
Inclusion Criteria:

* ● Age between 18 and 60 years.

  * Willingness and ability to fully understand the content and scope of the experiment and comply with its instructions.
  * Have signed the informed consent.

Exclusion Criteria:

* ● Pregnancy.

  * Ongoing chronic pain or neuromuscular disorder, or any Desis that effect the nociceptive system and not allowed to be evaluated in normal Condition
  * History of addictive behavior, defined as abuse of alcohol, cannabis, opioids, or other drugs.
  * History of heat sensitivity disorders.
  * History of mental illness.
  * Presence of fever, tuberculosis, malignant tumors, infectious processes, acute inflammatory processes
  * Implantation of pacemakers or metal prostheses.
  * Use of analgesics within 24 hours prior to participation in the experiment.
  * Lack of sleep (< 6 hours) the night before the experiment.
  * High alcohol intake the evening before the experiment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Latency and amplitude of the evoked potentials induce by pinprick stimuli | 2 hours during each experimental setting
  Latency (ms) and amplitude (mv) of the evoked potentials after pinprick stimulation
Latency and amplitude of the evoked potentials induce by RF | 2 hours during each experimental setting
  Latency (ms) and amplitude (mv) of the evoked potentials after RF

SECONDARY OUTCOMES:
Changes in responses to somatosensory stimuli with Pinprick thresholds | after each pinprick stimulation
  Intensity of pinprick sensation measure using a Numerical Scale Rating ranging from 0 no sensation to 100 most painful sensation.
Conduction velocity in radiofrequency stimuli | 10 minutes at the end of the RF setting
  Conduction speed of the stimuli in the leg and arm (ms)

CONTACTS AND LOCATIONS:
Locations (1):
- Facutlad de ingenieria UNER, Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iannetti GD, Baumgartner U, Tracey I, Treede RD, Magerl W. Pinprick-evoked brain potentials: a novel tool to assess central sensitization of nociceptive pathways in humans. J Neurophysiol. 2013 Sep;110(5):1107-16. doi: 10.1152/jn.00774.2012. Epub 2013 May 15. PMID 23678019
- [Background] Backonja MM, Walk D, Edwards RR, Sehgal N, Moeller-Bertram T, Wasan A, Irving G, Argoff C, Wallace M. Quantitative sensory testing in measurement of neuropathic pain phenomena and other sensory abnormalities. Clin J Pain. 2009 Sep;25(7):641-7. doi: 10.1097/AJP.0b013e3181a68c7e. PMID 19692807
- [Background] van den Broeke EN, Lambert J, Huang G, Mouraux A. Central Sensitization of Mechanical Nociceptive Pathways Is Associated with a Long-Lasting Increase of Pinprick-Evoked Brain Potentials. Front Hum Neurosci. 2016 Oct 20;10:531. doi: 10.3389/fnhum.2016.00531. eCollection 2016. PMID 27812331
- [Background] Vuilleumier PH, Biurrun Manresa JA, Ghamri Y, Mlekusch S, Siegenthaler A, Arendt-Nielsen L, Curatolo M. Reliability of Quantitative Sensory Tests in a Low Back Pain Population. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):665-73. doi: 10.1097/AAP.0000000000000289. PMID 26222349